CLINICAL TRIAL: NCT03402399
Title: Defining the Molecular Risk in Israeli Patients With Secondary Compared to Primary Myelofibrosis
Acronym: MRMF01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0124-17
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Myelofibrosis, Primary; Myelofibrosis, Post PV; Myelofibrosis, Post ET
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Myelofibrosis (Other): Blood test
  Interventions: Other: Molecular analysis
- Secondary Myelofibrosis (Other): Blood test
  Interventions: Other: Molecular analysis

INTERVENTIONS:
Other: Molecular analysis — Blood test

SUMMARY:
The aim of the study is to determine the rate of HMR mutations in PMF and secondary MF (post PV/ET) subjects, and correlate the rate of mutations with clinical features as known prognostic scores.

DETAILED DESCRIPTION:
Main inclusion criteria:

1. Diagnosis of PMF, post PV MF or post ET MF according to the WHO 2008 classification
2. Age ≥ 18 years
3. Concurrent participation in clinical trials will be allowed.

Efficacy assessments will be evaluated by: HMR mutations rate, specific HMR mutations, disease duration, presence of splenomegaly, cytogenetic risk, DIPPS, IPSS, ET survival score and PV survival score.

The primary efficacy parameter to be assessed will be HMR mutation rate.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PMF, post PV MF or post ET MF according to the WHO 2008 classification
2. Age . 18 years
3. Patient is willing and capable of giving a written informed consent.
4. Concurrent participation in clinical trials will be allowed

Exclusion Criteria:

1. Unwilling or unable to provide informed consent
2. Prefibrotic MF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2017-12-10 (Actual); Primary Completion 2019-12-09 (Estimated); Study Completion 2020-12-09 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with one or more HMR mutations in primary compared to secondary (post PV/ET) MF | Baseline
  Proportions of patients with HMR mutations in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Maya Koren-Michowitz, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No